CLINICAL TRIAL: NCT03654066
Title: Prospective Single-Blinded Randomized Controlled Trial Comparing Botox or Botox With Esophageal Dilation in Patients With Achalasia
Brief Title: Botox or Botox With Esophageal Dilation in Patients With Achalasia
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Dhyanesh Patel, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181420
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Botulinum Toxins, Type A; Patient Reported Outcome Measures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Botulinum toxin (Active Comparator): A one time dose of Botulinum toxin (Botox) is injected into the muscle of the LES leading to blockage of acetylcholine release from nerve endings resulting in increased relaxation.
  Interventions: Drug: Botulinum toxin type A; Other: Patient reported outcomes; Diagnostic Test: Barium esophagram
- Botulinum toxin and dilation (Active Comparator): A one time dose of Botulinum toxin (Botox) is injected into the muscle of the LES leading to blockage of acetylcholine release from nerve endings resulting in increased relaxation. Subjects will also undergo distal esophageal dilation using a 20mm through the scope balloon positioned across the LES.
  Interventions: Drug: Botulinum toxin type A; Device: Endoscope balloon dilator; Other: Patient reported outcomes; Diagnostic Test: Barium esophagram

INTERVENTIONS:
Drug: Botulinum toxin type A — Botox injection in the LES
  Other Names: Botox
Device: Endoscope balloon dilator — Distal esophageal dilation
  Arms: Botulinum toxin and dilation
Other: Patient reported outcomes — Subjects will complete two patient reported outcome measures (Eckardt and MADS).
Diagnostic Test: Barium esophagram — Assess for radiologic severity of achalasia with barium column height measured 1 minute and 5 minutes after upright ingestion of barium

SUMMARY:
Achalasia is a rare esophageal motility disorder. Treatment of achalasia is aimed toward palliation of symptoms. These include botox injections to the lower esophageal sphincter (LES), pneumatic dilation, surgical myotomy, and per-oral endoscopic myotomy (POEM). Botox injections are frequently used for patients that have significant comorbidities. The primary aim of this study is to assess symptomatic response of patient with achalasia to esophageal dilation and botox injection to the LES compared to standard therapy of only botox injection.

ELIGIBILITY:
Inclusion Criteria:

* Adults with known diagnosis of achalasia who are NOT candidates for definitive therapy with pneumatic dilation, surgical myotomy, or POEM
* Patient undergoing routine care upper endoscopy for achalasia

Exclusion Criteria:

* Less than 18 years old
* Previous surgery for reflux or peptic ulcer disease
* Significant medical conditions possibly placing subjects at risk to undergo endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
dysphagia score | 12 months
  Dysphagia score as measured by patient reported outcomes will be used to compare the two groups. The scale runs from 0 (no symptoms) to 100 (severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Dhyanesh Patel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee, United States